CLINICAL TRIAL: NCT02641535
Title: Evaluating the Physiological Strain Induced by a BC Membrane Protective Garment Under Exercise-heat Stress Compared to a Protective Coverall
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SHEBA-15-2689-OF-CTIL
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Physiological Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- research arm (Experimental): 12 healthy volunteers from the border guard of the police forces will participate in this study. The subjects will undergo 4 experiment days:
  1. Recruitment , medical examination and VO2max test.
  2. Acclimatization day by performing moderate exercise protocol under hot and humid climate.
  3.2 days of performing moderate exercise under hot and humid conditions protocol, each day dressed with different protective garment:
  1. Protective garment in current use + NBC mask.
  2. The new BC membrane protective garment + NBC mask
  Interventions: Other: exercise under hot and humid conditions protocol; Device: BC membrane protective garment; Device: NBC mask

INTERVENTIONS:
Other: exercise under hot and humid conditions protocol — acclimatization day protocol: 2 hour effort performed in a climatic chamber, which include walk on a treadmill at 5 Km/h on a 2% incline under heat conditions (40 deg. centigrade & 40% RH) Core (rectal) and skin temperature and heart rate will be monitored continuously
  experiment days (2 days): 2 hour effort (2 cycles of: 50 min walk and 10 min rest-sitting) performed in a climatic chamber, which include walk on a treadmill at 5 Km/h on a 2% incline under heat conditions (35 deg. centigrade & 60% RH) Core (rectal) and skin temperature and heart rate will be monitored continuously.
Device: BC membrane protective garment
Device: NBC mask

SUMMARY:
Israel ministry of defense is examining a new BC membrane protective garment of BLAUER company constructed with GORE CHEMPAK fabric for the border guard of the police forces. The goal of this research is to perform a comparative experiment in order to evaluate the physiological strain induced by the new protective garment under exercise-heat stress conditions, compared to protective garment in current use.

DETAILED DESCRIPTION:
In order to physiologically evaluate a new BC membrane protective garment for the Israeli police use under exercise-heat stress conditions, 12 healthy volunteers from the border guard will participate in this study.

The subjects will undergo 4 experiment days: Recruitment day, one day of acclimatization to heat, and 2 days of performing experiment protocol, each day dressed with different protective garment (Protective garment in current use + NBC mask, new BC membrane protective garment + NBC mask).

Core (rectal) and skin temperature and heart rate will be monitored continuously, liquid balance will be recorded.the physiological heat strain will be assessed and compared between the different protective garments.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40 years.
* Healthy civilian volunteers.
* Without known medical illness or medication use.

Exclusion Criteria:

* The existence or suspicion of existing cardiac or respiratory disease.
* Hypertension.
* Diabetes.
* Psychiatric condition.
* Any muscles or skeleton condition.
* Any hormonal disease or any other chronic illness that may inhibit participation in the experiment.
* Infectious disease 3 days prior to the experiment.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
physiological strain (composite) | 3 days for each participant
  The physiological strain will be determined by body core temperature and heart rate of the subjects during experiment days with protocol of exercise under heat stress conditions.

SECONDARY OUTCOMES:
Rectal temperature | 3 days for each participant
  The rectal temperature will be monitored by a rectal thermistor (YSI-401) inserted 10 cm past the anal sphincter.
Skin temperature | 3 days for each participant
  The skin temperature will be monitored by skin thermistors located at 3 sites (chest, arm and leg).
Heart rate | 4 days for each participant
  The heart rate will be monitored using a wearable heart rate monitor (Polar® sensor and heart rate monitor watch).
Sweat rate (composite) | 3 days for each participant
  Sweat rate will be calculated from the patients' body weight and fluid balance.

CONTACTS AND LOCATIONS:
Overall Officials: Ofir Frenkel, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Ramat- Gan, Israel